CLINICAL TRIAL: NCT00888875
Title: Is Fiberoptic Intubation Through the I-gel™ Equal to Fiberoptic Intubation Through the Intubating Laryngeal Mask (Fastrach)™ ?
Brief Title: ILMA Fastrach Versus I-gel for Fiberoptic Tracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fast igel1
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Tracheal Intubation
Keywords: i-gel; Fastrach; intubation; fiberoptic; difficult airway; Patients undergoing elective surgery requiring tracheal intubation; Presenting at least one sign of difficult intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Computer randomized insertion of the i-gel. Intubation fiberoptically of a tracheal tube
  Interventions: Device: i-gel
- 2 (Active Comparator): Computer randomized insertion of the i-gel. Intubation fiberoptically of a tracheal tube
  Interventions: Device: ILMA

INTERVENTIONS:
Device: i-gel — insertion after induction of anaesthesia. Afterwards, intubation over the device fiberoptically
  Arms: 1
Device: ILMA — Insertion after Induction. Insertion of tracheal tube over device
  Arms: 2

SUMMARY:
We evaluate feasibility of fiberoptic intubation through the "ILMA Fastrach" vs the "i-gel". Both are airway devices to be introduced in the mouth we the possibility to ventilate the patient and furthermore to be a guide to introduce a tracheal tube. We first insert either the ILMA or the i-gel. In a second step, we will introduce a tube through the device, all guided visually through a fiberoptic tool which works as a railroad for the tracheal tube.

DETAILED DESCRIPTION:
The ILMA Fastrach™ is a widely accepted and intensively investigated supraglottic airway device that is inserted blindly. It may be used to facilitate intubation and secure the airway in routine practice, in difficult airway scenarios or in emergency situations. Endotracheal tube insertion may be blind or fiberoptic scope guided, the latter raises the success rate. The i-gel™ is a newly developed supraglottic airway device and is also introduced blindly. Insertion of an endotracheal tube may be blind or fiberoptically guided.

So far, prospective randomized controlled trials comparing their performance are not yet published. There are case reports about intubating over the i-gel.

In this prospective, randomized, controlled trial, we are going to evaluate the performance of intubation through both devices. In 250 patients undergoing elective surgery, we will place either the ILMA or the i-gel according to randomization and then intubate with the help of a fiberoptic scope, using the specific ILMA tracheal tube or a normal tracheal tube for the i-gel. In order to remove the supraglottic airway devices, we will use the ILMA stabilizer rod.

ELIGIBILITY:
Inclusion Criteria:

* elective operation with intubation
* ASA I-IV
* speaks German
* at least one predictor for difficult intubation

Exclusion Criteria:

* weight <30kg
* Risk Aspiration
* Risk bleeding orally
* known or highly suspected difficult mask ventilation
* Mouth opening < 20mm

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2008-07; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
successful intubation attempt with ventilation of both lungs | during intervention

SECONDARY OUTCOMES:
insertion of supraglottic airway devices, the time to intubate, airway device leak pressure, adverse events and postoperative side effects | during intervention and first 24hours after operation
simulated blind intubation in both groups | during intervention

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, M.D., Study Director — Department of Anesthesia, University Hospital Berne, Switzerland
Locations (1):
- University Hospital, Bern, Canton of Bern, Switzerland